CLINICAL TRIAL: NCT07071285
Title: Applying Interactive E-books on Breastfeeding to Enhance Nursing Students' Learning Motivation and Effectiveness in Breastfeeding Education
Brief Title: Applying Interactive E-books on Breastfeeding to Enhance Nursing Students' Learning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ting-Shan Chang, Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUH114-REC3-125
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Nursing Education Research; Nursing Students; Breastfeeding Education
Keywords: e-book; nursing education; learning motivation; Breastfeeding Education; Nursing Students

STUDY DESIGN:
Intervention Model Description: The study design will adopt a randomized controlled trial with repeated measures. A 60-minute intervention has been developed.Block randomization stratified by gender will be used, and eligible participants will be randomly assigned to either the experimental or control group in a 1:1 ratio using Random Allocation Software.Research assistants will code group assignments ("Group 1" and "Group 2") according to the randomization list, place the assignments into opaque sealed envelopes, and arrange them sequentially.On the day of the study, envelopes will be distributed in the order participants submit their consent forms. Participants will open the envelope themselves to learn their group assignment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-book (Experimental): Breastfeeding eBook learning mode.
  Interventions: Behavioral: E-Book
- face-to-face teaching (Active Comparator): face-to-face teaching of breastfeeding
  Interventions: Behavioral: face-to-face teaching

INTERVENTIONS:
Behavioral: E-Book — Breastfeeding eBook learning mode.
  Arms: E-book
Behavioral: face-to-face teaching — face-to-face teaching of breastfeeding
  Arms: face-to-face teaching

SUMMARY:
This study aims to explore the impact of interactive breastfeeding e-books on nursing students' breastfeeding learning outcomes. The subjects are third-year nursing students from a university in central Taiwan. A randomized controlled design will be adopted. The experimental group will use interactive breastfeeding e-books for learning, while the control group will use traditional face-to-face courses to evaluate the changes in students' breastfeeding knowledge, skills, and learning motivation. The expected results can provide a reference for innovative teaching models in nursing education and promote the future clinical promotion of breastfeeding.

DETAILED DESCRIPTION:
Breastfeeding is widely considered to be the best source of nutrition for infants, helping to reduce infant morbidity and mortality, reduce the risk of infection and chronic diseases, and promote intellectual development. However, in current nursing education, how to effectively improve students' knowledge and skills of breastfeeding has yet to be developed. Common traditional face-to-face courses are limited by time and venue, which requires students to re-adapt and learn when entering the clinical internship stage, affecting learning efficiency and clinical application. In addition, male students may find it challenging to learn breastfeeding due to gender factors.

With the rapid development of information technology, e-books and multimedia interactive teaching materials have been proven to improve learning motivation and effectiveness, promote individualized learning experience, and enhance problem solving and creative thinking. Through animation, sound effects, pictures, and game quizzes, it can effectively help students master professional knowledge and overcome the limitations of traditional teaching.

This study adopts a randomized controlled experimental design and is expected to recruit 100 third-year nursing students from a university in central Taiwan, divided into an experimental group and a control group. The experimental group studied with an interactive breastfeeding e-book, and the control group took a traditional face-to-face course. Data were collected through a structured questionnaire, and changes in breastfeeding knowledge, skill acquisition, and learning motivation were analyzed using descriptive and inferential statistics. The expected results showed that the interactive e-book not only significantly improved students' learning outcomes, but also helped overcome gender restrictions, enhance learning motivation, promote future clinical promotion of breastfeeding, and serve as an important reference for innovative nursing education models.

ELIGIBILITY:
Inclusion Criteria:

1. It is expected to include 100 people.
2. Age 20 to 30 years old.
3. A third-year nursing student.
4. Studying obstetrics and gynecology nursing this semester.
5. Agree to participate in this study and sign the research consent form.

Exclusion Criteria:

1 .Students who are planning to take a leave of absence at the time of data collection.

2.Students who have not taken obstetrics and gynecology nursing this semester or have taken it in the past.

3.Students who are unable to use 3C products.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Knowledge Questionnaire | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  This questionnaire consists of 10 multiple-choice questions. Each correct answer is scored 10 points, and each incorrect answer is scored 0 points, yielding a total score range of 0-100. The questions were self-developed in the form of clinical scenario-based multiple-choice items, focusing on the benefits of breastfeeding, breastfeeding positions, breast milk storage methods, breast milk expression (hand expression), and nursing interventions to maintain milk supply.
Breastfeeding Skills Assessment Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  Breastfeeding skills were assessed using a "Breastfeeding Skills Assessment Scale," which includes 20 steps such as hand hygiene before procedures, self-introduction, patient identification, ensuring privacy, explaining the purpose and process, breastfeeding positions, and hand expression techniques. Each step is scored as follows: completely correct = 5 points, partially correct = 3 points, and incorrect = 0 points. The total score ranges from 0-100, with higher scores indicating better application of breastfeeding skills.
Breastfeeding Self-Efficacy Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  Breastfeeding self-efficacy was evaluated using a 10-item Breastfeeding Self-Efficacy Scale. Each item is rated on a 4-point Likert scale, where 1 = not at all capable and 4 = expert level. The total score ranges from 10 to 40, with higher scores indicating greater self-efficacy in performing breastfeeding skills.
ARCS-Based Learning Motivation Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  The scale assesses learners' motivation toward the educational materials across four dimensions: Attention (12 items), Relevance (9 items), Confidence (9 items), and Satisfaction (6 items), for a total of 36 items. Responses are rated on a 5-point Likert scale, ranging from 5 ("Strongly Agree") to 1 ("Strongly Disagree"). The total score ranges from 36 to 180 points, with higher scores indicating stronger learning motivation.
Critical Thinking Disposition Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  This scale consists of 20 items and adopts a 6-point Likert scoring method: 1 (Never), 2 (Almost Never), 3 (Rarely), 4 (Sometimes), 5 (Often), and 6 (Always). It measures critical thinking disposition, which refers to an individual's tendency to engage in systematic analysis, maintain an open-minded attitude with empathy, and possess a wise curiosity for questioning, integration, and reflection, all of which facilitate critical thinking processes.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan, Taiwan